CLINICAL TRIAL: NCT06307938
Title: Circulating Tumor DNA in Patients Summoned for Colonoscopy; - a Liquid Biopsy for Detection, Characterization, Individualized Treatment and Follow-up of Colorectal Cancer
Acronym: CoLiQ
Status: Recruiting | Type: Observational
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 619020
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer; Colorectal Adenoma
Keywords: Biomarker; Liquid biopsy; ctDNA
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: liquid biopsy — based on a panel of circulating tumor DNA markers

SUMMARY:
CoLiQ is a clinical study designed to evaluate the clinical usefulness of circulating tumor DNA (ctDNA) markers found in blood, as a liquid biopsy for diagnosis, prognosis and follow-up of colorectal cancer. The main questions it aims to answer are: 1) Can a panel of ctDNA markers identify CRC patients among the other patients summoned for colonoscopy? and 2) Does the type, number and level of ctDNA markers vary with the subtype and clinical course of CRC? Participants will be asked to answer a questionnaire and give a blood sample at inclusion. In addition, patients with CRC will be asked to give an extra test tube at their routine treatment and follow-up blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old summoned for colonoscopy
* Patient able to understand and sign written informed consent

Exclusion Criteria:

* Patient < 18 years old
* Patient unable to understand or give written informed consent
* Patient unlikely to comply with the protocol (e.g. uncooperative attitude, inability to return for subsequent visits) and/or otherwise considered by the investigator as unlikely to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients summoned for colonoscopy at their local public hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer | evaluated within 3 months after colonoscopy
  Number of patients with colorectal cancer at histology following colonoscopy
Colorectal adenoma | evaluated within 3 months after colonoscopy
  Number of patients with colorectal adenoma at histology following colonoscopy
Inflammatory bowel disease | evaluated within 3 months after colonoscopy
  Number of patients with inflammatory bowel disease at histology following colonoscopy

SECONDARY OUTCOMES:
Recurrence | Within 5 years following treatment with curative intent for colorectal cancer
  Recurrence of colorectal cancer among patients treated curatively.
Death | Within 5 years following diagnosis of colorectal cancer
  Death among patients with colorectal cancer
Treatment response | Within the 5 years following diagnosis of colorectal cancer
  Treatment response among colorectal cancer patients as measured by todays standards of follow-up (CEA, CT-scans, colonoscopy)

CONTACTS AND LOCATIONS:
Locations (1):
- Nord-Trøndelag Hospital Trust, Levanger, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.hnt.no/kliniske-studier/coliq--fra-koloskopi-til-flytende-biopsi/